CLINICAL TRIAL: NCT03756272
Title: Short-term Efficacy of Stellate Ganglion Block to Reduce Hot Flushes
Brief Title: Stellate Ganglion Block to Reduce Hot Flushes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL54465.091.15
Record Dates: First submitted 2017-09-22; First posted 2018-11-28 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hot Flash; Stellate Ganglion Block; Postmenopausal; Hot Flushes
MeSH Terms: conditions — Hot Flashes | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: In this study patient and outcome assessor are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate ganglion bupivacaine block (Experimental): Nervus Sympathicus block. Stellate ganglion anaesthetic block in which 7 ml of 0.5% bupivacaine will be injected next to the stellate ganglion
  Interventions: Procedure: Bupivacaine block
- Placebo ganglion block (Placebo Comparator): Sham Nervus Sympathicus block. Stellate ganglion sham anaesthetic block using 7 ml of 0.9 % natrium chloride (NaCl)
  Interventions: Procedure: Placebo ganglion block

INTERVENTIONS:
Procedure: Bupivacaine block — stellate ganglion bupivacaine injection
  Other Names: Stellate ganglion Block
  Arms: Stellate ganglion bupivacaine block
Procedure: Placebo ganglion block — stellate ganglion sodium chloride injection
  Other Names: stellate ganglion natrium chloride 0.9% injection
  Arms: Placebo ganglion block

SUMMARY:
To assess the short-term efficacy of stellate ganglion block on hot flush reduction versus sham procedure

DETAILED DESCRIPTION:
Hot flushes are the most common symptom of menopause for which postmenopausal (PMP) women seek medical help, in 20% of PMP women hot flushes can persist for up to 15 years.

A possible treatment for hot flushes is stellate ganglion block (SGB), used as a means to interrupt parts of the sympathetic nervous system involved in temperature regulation.

Single centre randomized double blind placebo controlled intervention study Study period of 6 months in which patients will fill out on set time points 5 questionnaires regarding quality of life and keep a diary on hot flush frequency and severity during1 week on the same time points.

Study population:

Postmenopausal women aged 30-70 years old with no other causes of flushing present. Intervention (if applicable) Intervention: Stellate ganglion block versus sham procedure

Follow up with questionnaires during 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age: 30-70 years
* Mean daily flush frequency of 10 or more and a hot flush score of 15 or more
* Absence of any non-menopausal cause of flushing
* Post-menopause amenorrhea for more than 1 year in healthy postmenopausal women
* In case of breast cancer or ovariectomy induced menopause: ovariectomy for > 6 months. Adjuvant therapy with estrogen-receptor blocker or an aromatase inhibitor.

Exclusion Criteria:

* Use of medication that affects flushing:oestrogens, progestogens, clonidine, naloxone, paroxetine, fluoxetine, venlafaxine, gabapentin, luteïniserend hormone releasing hormones receptor antagonist
* Receiving chemotherapy of radiotherapy
* Active psychiatric disease
* Active concurrent disease
* Allergic reactions against local anesthetics of the 'amide' type or contrast media.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-04-28 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Hot Flush score | Baseline, 4, and 8 weeks
  Hot flush score as measured by a hot flush diary in which for each hot flush the severity is noted for one week. Severity of every flush is given on a 1-4 scale (1 is mild, 2 medium, 3 severe, and 4 is very severe)

SECONDARY OUTCOMES:
Quality of sleep | Baseline, 4, and 8 weeks
  Pittsburgh Sleep Quality Index: developed to discriminate between good and poor sleep quality. It consists of 19 individual items, creating seven components of sleep (sleep onset latency, sleep duration, sleep efficiency, sleep quality, sleep disturbances,medication, and day-time dysfunction). Each of those seven components is scored from 0 to 3. The sum of the individual scores forms the global score (0-21) of the PSQI. Lower global scores denote high sleep quality, whereas a score greater than 5 is considered poor sleep quality
Sleepiness | Baseline, 4, and 8 weeks
  Epworth Sleepiness Scale. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The reference range of 'normal' ESS scores is zero to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Willem Kallewaard, MD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate hospital, Arnhem, Netherlands